CLINICAL TRIAL: NCT00602069
Title: Treatment of PTSD in Recently Battered Women Living in Shelters
Brief Title: Cognitive Behavioral Therapy for Treating Recently Abused Women With Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Akron (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Summa Health System (Other); Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH080786 (NIH); R34MH080786 (NIH); DATR AD-TS
Record Dates: First submitted 2008-01-18; First posted 2008-01-28 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Post-Traumatic Stress Disorder; Battered Women
Keywords: PTSD; Intimate Partner Violence; Cognitive Behavioral Therapy; Empowerment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Empowerment | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive cognitive behavioral therapy through the Helping to Overcome PTSD through Empowerment program
  Interventions: Behavioral: Helping to Overcome PTSD through Empowerment (HOPE)
- 2 (Active Comparator): Participants will receive standard shelter services
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Helping to Overcome PTSD through Empowerment (HOPE) — HOPE includes a maximum of 16 sessions of cognitive behavioral therapy. The sessions will emphasize stabilization and empowerment, both of which are identified as important goals by the theoretical and empirical literature on abused women and PTSD.
  Other Names: HOPE
  Arms: 1
Behavioral: Treatment as usual — Treatment as usual includes standard shelter services for abused women.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a brief cognitive behavioral treatment, Helping to Overcome PTSD through Empowerment, in treating abused women with post-traumatic stress disorder who are living in shelters.

DETAILED DESCRIPTION:
Intimate partner violence is a serious social problem with potentially severe mental health and functional consequences consistent with post-traumatic stress disorder (PTSD). Shelters provide an important resource for abused women in that they offer emergency shelter, support, and access to community resources that can aid in establishing long-term safety for women and their children. However, recent research suggests that symptoms of PTSD can compromise abused women's ability to access and effectively use these resources, emphasizing the importance of initiating treatment for PTSD. Despite the fact that on an annual basis 300,000 battered women and children access shelter services, virtually no research has investigated treatment of PTSD in sheltered abused women. A woman's entry into a shelter seems to be a prime time to begin any necessary psychological treatment. Helping to Overcome PTSD through Empowerment (HOPE), a brief cognitive behavioral treatment that emphasizes stabilization and empowerment of women, may help in treating abused women with PTSD. This study will evaluate the effectiveness of HOPE in treating abused women with PTSD who are in shelters.

Participation in this single-blind study will begin during a woman's shelter stay and will end 8 months after she completes the shelter treatment period. All potential participants will first undergo an initial interview, which will include questions about their abusive relationships, emotional difficulties, stressful events, and other previous treatments. Participants invited to continue with the study will be randomly assigned to the HOPE program or to shelter treatment as usual. Participants assigned to the HOPE program will participate in a maximum of 16 counseling sessions, with up to 10 of these sessions taking place while they are at the shelter. During these sessions, participants will learn skills to help manage emotional difficulties and ways to deal with their abusive relationships. Participants will attend two 60- to 90-minute sessions each week until they complete of the 10 shelter-based counseling sessions or depart from the shelter. Counseling sessions will continue at St. Thomas Hospital or other agreed-upon location twice per week during the first 8 weeks after departure from the shelter. All participants will repeat the initial interview and/or questionnaire at various times during and after the shelter stay, for a total of eight assessments. The final interview assessment will occur 6 months after participants complete the counseling sessions.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for PTSD or subthreshold PTSD
* Resident of a battered women's shelter
* Abused in the month prior to study entry

Exclusion Criteria:

* Significant suicidal ideation or risk
* Current psychotic symptoms
* Current alcohol or drug dependence
* Lifetime history of bipolar disorder
* Concurrent psychosocial treatment
* Any change in medication in the month prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity | Measured at Month 8

SECONDARY OUTCOMES:
Effective use of resources | Measured at Month 8
Resource loss | Measured at Month 8
Depression | Measured at Month 8
Social functioning | Measured at Month 8
Revictimization | Measured at Month 8

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Johnson, PhD, Principal Investigator — Summa Health System
Locations (1):
- University of Akron, Akron, Ohio, United States

REFERENCES:
- [Background] Johnson DM, Zlotnick C. A cognitive-behavioral treatment for battered women with PTSD in shelters: findings from a pilot study. J Trauma Stress. 2006 Aug;19(4):559-64. doi: 10.1002/jts.20148. PMID 16929512
- [Derived] Johnson DM, Johnson NL, Perez SK, Palmieri PA, Zlotnick C. Comparison of Adding Treatment of PTSD During and After Shelter Stay to Standard Care in Residents of Battered Women's Shelters: Results of a Randomized Clinical Trial. J Trauma Stress. 2016 Aug;29(4):365-73. doi: 10.1002/jts.22117. Epub 2016 Jul 26. PMID 27459503